CLINICAL TRIAL: NCT04205058
Title: Coffee After Pancreatic Surgery - a Randomised, Single Blinded, Placebo-controlled Trial
Brief Title: Coffee After Pancreatic Surgery
Acronym: COPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2296CESC
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Ileus; Postoperative Complications; Bowel Dysfunction; Pancreatic Diseases
Keywords: Randomised clinical trial; Pancreatic surgery
MeSH Terms: conditions — Postoperative Complications; Intestinal Diseases; Pancreatic Diseases | interventions — Drinking Water

STUDY DESIGN:
Intervention Model Description: randomised placebo-controlled single blinded trial
Who Masked: Participant
Masking Description: Participants are masked about the type of coffee administrated (standard coffee versus caffeine-free coffee). Masking about administration of hot water is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard coffee (Experimental): Hot standard coffee with caffeine (one 30 mL espresso cup twice a day, from postoperative day one to first bowel movement or postoperative day three).
  Interventions: Dietary Supplement: Standard coffee
- caffeine-free coffee (Placebo Comparator): Hot caffeine-free coffee (one 30 mL espresso cup twice a day, from postoperative day one to first bowel movement or postoperative day three).
  Interventions: Dietary Supplement: Caffeine-free coffee
- water (Sham Comparator): Hot water (one 30 mL espresso cup twice a day, from postoperative day one to first bowel movement or postoperative day three).
  Interventions: Dietary Supplement: Drinking water

INTERVENTIONS:
Dietary Supplement: Standard coffee — One 30 mL espresso cup administered twice a day (08.00 a.m. and 02.00 p.m.).
  Arms: standard coffee
Dietary Supplement: Caffeine-free coffee — One 30 mL espresso cup administered twice a day (08.00 a.m. and 02.00 p.m.).
  Arms: caffeine-free coffee
Dietary Supplement: Drinking water — One 30 mL espresso cup administered twice a day (08.00 a.m. and 02.00 p.m.).
  Arms: water

SUMMARY:
Postoperative ileus is a common complication after major abdominal surgery. A positive effect of coffee to bowel movement has been described after colorectal and gynecologic interventions. The objective of this randomised controlled trial is to investigate whether the implementation of a fast track protocol with early coffee consumption accelerates the recovery of bowel function after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a common disorder after major abdominal surgery, affecting up to 40% of patients undergoing laparotomy. POI is described as the time between surgery and the first passage of flatus and/or stool and tolerance of oral diet. It could be recognised as postoperative complication when is defined as two or more of nausea/vomiting, inability to tolerate oral diet over 24 h, absence of flatus over 24 h, abdominal distention and radiologic confirmation on or after day 4 postoperatively without prior resolution. Multimodal approaches have been described to treat POI; among them, the early consumption of coffee showed a substantial benefit after colorectal and gynecologic surgery. The objective of this randomised placebo-controlled trial is to investigate whether early coffee consumption can accelerate the recovery of bowel function after open pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Elective open pancreaticoduodenectomy
* Age ≥ 18 years
* American Society Anesthesiologists (ASA) score ≤ 3
* Ability of the subject to understand aims and clinical consequences of the trial
* Written informed consent

Exclusion Criteria:

* American Society Anesthesiologists (ASA) score ≥ 4
* Need for early postoperative Intensive Care Unit care
* Need for naso-gastric tube on postoperative day one
* Intolerance to coffee
* Refuse to assume coffee
* Pregnancy
* Surgical procedures performed different from pancreaticoduodenectomy
* Impaired mental status or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-12-05 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
First Bowel Movement | 96 hours.
  Time to first bowel movement (expressed by hours from the time of surgical procedure ending).

SECONDARY OUTCOMES:
First Flatus | 96 hours
  Time to first flatus (expressed by hours from the time of surgical procedure ending).
Tolerance to solid food | 96 hours
  Time to tolerance to solid food (expressed by hours from the time of surgical procedure ending). Tolerance was defined as the ability to eat at least half of the solid food served by hospital staff.
Length of stay | 90 days
  Length of stay expressed by days from intervention to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassi, MD, Study Director — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassen K, Coolsen MM, Slim K, Carli F, de Aguilar-Nascimento JE, Schafer M, Parks RW, Fearon KC, Lobo DN, Demartines N, Braga M, Ljungqvist O, Dejong CH; ERAS(R) Society; European Society for Clinical Nutrition and Metabolism; International Association for Surgical Metabolism and Nutrition. Guidelines for perioperative care for pancreaticoduodenectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):817-30. doi: 10.1016/j.clnu.2012.08.011. Epub 2012 Sep 26. PMID 23079762
- [Background] Vather R, Trivedi S, Bissett I. Defining postoperative ileus: results of a systematic review and global survey. J Gastrointest Surg. 2013 May;17(5):962-72. doi: 10.1007/s11605-013-2148-y. Epub 2013 Feb 2. PMID 23377782
- [Background] Artinyan A, Nunoo-Mensah JW, Balasubramaniam S, Gauderman J, Essani R, Gonzalez-Ruiz C, Kaiser AM, Beart RW Jr. Prolonged postoperative ileus-definition, risk factors, and predictors after surgery. World J Surg. 2008 Jul;32(7):1495-500. doi: 10.1007/s00268-008-9491-2. PMID 18305994
- [Background] Story SK, Chamberlain RS. A comprehensive review of evidence-based strategies to prevent and treat postoperative ileus. Dig Surg. 2009;26(4):265-75. doi: 10.1159/000227765. Epub 2009 Jul 3. PMID 19590205
- [Background] Asgeirsson T, El-Badawi KI, Mahmood A, Barletta J, Luchtefeld M, Senagore AJ. Postoperative ileus: it costs more than you expect. J Am Coll Surg. 2010 Feb;210(2):228-31. doi: 10.1016/j.jamcollsurg.2009.09.028. Epub 2009 Nov 18. PMID 20113944
- [Background] Muller SA, Rahbari NN, Schneider F, Warschkow R, Simon T, von Frankenberg M, Bork U, Weitz J, Schmied BM, Buchler MW. Randomized clinical trial on the effect of coffee on postoperative ileus following elective colectomy. Br J Surg. 2012 Nov;99(11):1530-8. doi: 10.1002/bjs.8885. Epub 2012 Sep 14. PMID 22987303
- [Background] Dulskas A, Klimovskij M, Vitkauskiene M, Samalavicius NE. Effect of Coffee on the Length of Postoperative Ileus After Elective Laparoscopic Left-Sided Colectomy: A Randomized, Prospective Single-Center Study. Dis Colon Rectum. 2015 Nov;58(11):1064-9. doi: 10.1097/DCR.0000000000000449. PMID 26445179
- [Background] Gungorduk K, Ozdemir IA, Gungorduk O, Gulseren V, Gokcu M, Sanci M. Effects of coffee consumption on gut recovery after surgery of gynecological cancer patients: a randomized controlled trial. Am J Obstet Gynecol. 2017 Feb;216(2):145.e1-145.e7. doi: 10.1016/j.ajog.2016.10.019. Epub 2016 Oct 22. PMID 27780709
- [Background] Hasler-Gehrer S, Linecker M, Keerl A, Slieker J, Descloux A, Rosenberg R, Seifert B, Nocito A. Does Coffee Intake Reduce Postoperative Ileus After Laparoscopic Elective Colorectal Surgery? A Prospective, Randomized Controlled Study: The Coffee Study. Dis Colon Rectum. 2019 Aug;62(8):997-1004. doi: 10.1097/DCR.0000000000001405. PMID 30998528
- [Background] Bassi C, Molinari E, Malleo G, Crippa S, Butturini G, Salvia R, Talamini G, Pederzoli P. Early versus late drain removal after standard pancreatic resections: results of a prospective randomized trial. Ann Surg. 2010 Aug;252(2):207-14. doi: 10.1097/SLA.0b013e3181e61e88. PMID 20622661